CLINICAL TRIAL: NCT05026541
Title: Resilience to Sleep Deprivation and Changes in Sleep Architecture in Shoonya Meditators
Acronym: REST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021P000544
Record Dates: First submitted 2021-07-19; First posted 2021-08-30 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Sleep; Sleep Deprivation; Cognitive Change
Keywords: sleep; sleep disorder; sleep deprivation; Meditation; Shoonya meditation
MeSH Terms: conditions — Sleep Deprivation; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nap Practitioners (Sham Comparator): This is an observational arm of regular nappers. Individuals that take naps at least two times a week will be invited to undergo all of the study procedures for one weekend of data collection.
  Interventions: Behavioral: Nap Practitioners
- Shoonya Meditators (Active Comparator): This is intervention arm. Participants will learn and practice the fifteen minute shoonya meditation - described as a process of conscious non-doing- and shakti chalana kriya, which is a set of breathing exercises designed as a preparatory practice to shoonya meditation. Participants will practice shoonya meditation twice a day for two months. A weekend of data collection will happen at baseline and two months after they learn the practice.
  Interventions: Behavioral: Shoonya Meditation
- Control Meditators (No Intervention): Control subjects will be individuals that have learned the prerequisite meditation to Shoonya meditation. This meditation is called Shambhavi Mahamudra Kriya. Control subjects will not learn Shoonya meditation while they are participating in the study. One weekend of data collection will occur at baseline.

INTERVENTIONS:
Behavioral: Nap Practitioners — Regular nappers will be given a 30 minute nap opportunity to nap for as long as they please.
  Arms: Nap Practitioners
Behavioral: Shoonya Meditation — This is a 15 minute meditation, described as a process of conscious non-doing.
  Arms: Shoonya Meditators

SUMMARY:
This study aims to investigate the effect of a 15-minute meditation practice on sleep architecture and high-frequency Heart Rate Variability (HF-HRV), as well as cognitive performance after both a well-rested and sleep-deprived night.

DETAILED DESCRIPTION:
Sleep is physiologically important for memory consolidation, mood and hormonal regulation, and maintaining low levels of systemic inflammation. However, a substantial proportion of people are reported to regularly sleep less than the recommended 7-9 hours a night. Meditation may be a means to mitigate the negative effects of sleep deprivation, as many types of meditations are associated with increasing high-frequency heart rate variability (HF-HRV), which is an index of parasympathetic control of the heart. Greater parasympathetic drive may be associated with physiological buffering of the detrimental effects of sleep deprivation.

The investigators want to conduct a prospective cohort study where subjects are asked to learn and practice a 15-minute meditation (shoonya meditation) or continue their usual routine. Subjects will be asked to complete some cognitive tests before and after a night of sleep and a night of sleep deprivation. During the night of sleep, participants will undergo polysomnography recording for sleep architecture and quality.

The intervention group will be asked to undergo these same study procedures after 2 months of meditation practice. The control group, which continues their usual routine, will only undergo one visit.

ELIGIBILITY:
Inclusion Criteria:

1. Shoonya meditation program participants/individuals eligible to participate who are healthy adults of age 18 or older, and reside in the United States. Participants must be able and willing to travel to Boston.
2. Nap Group: Healthy adults of age 18 or older that reside in the United States, nap regularly (at least 3 times a week), and do not meditate regularly.

Exclusion Criteria:

1. History of any neurological condition (i.e. Parkinson's disease, Alzheimer's disease, Huntington's disease, brain tumors, brain surgery, or multiple sclerosis)
2. History of any psychiatric disorder, within last 5 years (i.e. anxiety, psychosis, posttraumatic stress disorder, attention deficit hyperactive disorder)
3. Current use of cognition enhancing medications
4. Active history (within the last 5 years) of alcohol or drug abuse (> 10 drinks per week)
5. History (within the last 5 years) of stroke/aneurysm
6. Recent history (< 3 months) of seizures
7. 60 years of age or older
8. History of Heart Attack and Ejection Fraction less than or equal to 30%
9. Pregnancy
10. Non-English speaking
11. History/Diagnosis of any sleep disorder
12. Consumption of 3 or more cups of coffee a day
13. Previously learned shoonya meditation (for the meditator groups)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Error frequency Change: Go-No Go Task | 2 months post learning meditation
  The primary outcome is the difference in number of commission and omission errors on the Go-No Go task. The difference in scores pre- and post-sleep deprivation will be analyzed between the control and intervention group.

SECONDARY OUTCOMES:
Reaction Time Change: Go-No Go | 2 months post learning meditation
  The difference in reaction times on the Go-No Go task. The difference in scores pre- and post-sleep deprivation will compared between the control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States

REFERENCES:
- [Background] Heyde I, Kiehn JT, Oster H. Mutual influence of sleep and circadian clocks on physiology and cognition. Free Radic Biol Med. 2018 May 1;119:8-16. doi: 10.1016/j.freeradbiomed.2017.11.003. Epub 2017 Nov 10. PMID 29132973
- [Background] Hirshkowitz M, Whiton K, Albert SM, Alessi C, Bruni O, DonCarlos L, Hazen N, Herman J, Katz ES, Kheirandish-Gozal L, Neubauer DN, O'Donnell AE, Ohayon M, Peever J, Rawding R, Sachdeva RC, Setters B, Vitiello MV, Ware JC, Adams Hillard PJ. National Sleep Foundation's sleep time duration recommendations: methodology and results summary. Sleep Health. 2015 Mar;1(1):40-43. doi: 10.1016/j.sleh.2014.12.010. Epub 2015 Jan 8. PMID 29073412
- [Background] Ben Simon E, Rossi A, Harvey AG, Walker MP. Overanxious and underslept. Nat Hum Behav. 2020 Jan;4(1):100-110. doi: 10.1038/s41562-019-0754-8. Epub 2019 Nov 4. PMID 31685950
- [Background] Krause AJ, Simon EB, Mander BA, Greer SM, Saletin JM, Goldstein-Piekarski AN, Walker MP. The sleep-deprived human brain. Nat Rev Neurosci. 2017 Jul;18(7):404-418. doi: 10.1038/nrn.2017.55. Epub 2017 May 18. PMID 28515433
- [Background] Tang YY, Holzel BK, Posner MI. The neuroscience of mindfulness meditation. Nat Rev Neurosci. 2015 Apr;16(4):213-25. doi: 10.1038/nrn3916. Epub 2015 Mar 18. PMID 25783612
- [Background] Braboszcz C, Cahn BR, Levy J, Fernandez M, Delorme A. Increased Gamma Brainwave Amplitude Compared to Control in Three Different Meditation Traditions. PLoS One. 2017 Jan 24;12(1):e0170647. doi: 10.1371/journal.pone.0170647. eCollection 2017. PMID 28118405
- [Background] Kaul P, Passafiume J, Sargent CR, O'Hara BF. Meditation acutely improves psychomotor vigilance, and may decrease sleep need. Behav Brain Funct. 2010 Jul 29;6:47. doi: 10.1186/1744-9081-6-47. PMID 20670413
- [Background] Maruthai N, Nagendra RP, Sasidharan A, Srikumar S, Datta K, Uchida S, Kutty BM. Senior Vipassana Meditation practitioners exhibit distinct REM sleep organization from that of novice meditators and healthy controls. Int Rev Psychiatry. 2016 Jun;28(3):279-87. doi: 10.3109/09540261.2016.1159949. Epub 2016 Apr 8. PMID 27055575
- [Background] Killgore WD. Effects of sleep deprivation on cognition. Prog Brain Res. 2010;185:105-29. doi: 10.1016/B978-0-444-53702-7.00007-5. PMID 21075236
- [Background] Thayer JF, Lane RD. Claude Bernard and the heart-brain connection: further elaboration of a model of neurovisceral integration. Neurosci Biobehav Rev. 2009 Feb;33(2):81-8. doi: 10.1016/j.neubiorev.2008.08.004. Epub 2008 Aug 13. PMID 18771686
- [Background] Lischke A, Lemke D, Neubert J, Hamm AO, Lotze M. Inter-individual differences in heart rate variability are associated with inter-individual differences in mind-reading. Sci Rep. 2017 Sep 14;7(1):11557. doi: 10.1038/s41598-017-11290-1. PMID 28912591
- [Background] Kong SDX, Hoyos CM, Phillips CL, McKinnon AC, Lin P, Duffy SL, Mowszowski L, LaMonica HM, Grunstein RR, Naismith SL, Gordon CJ. Altered heart rate variability during sleep in mild cognitive impairment. Sleep. 2021 Apr 9;44(4):zsaa232. doi: 10.1093/sleep/zsaa232. PMID 33306103
- [Background] Libby DJ, Worhunsky PD, Pilver CE, Brewer JA. Meditation-induced changes in high-frequency heart rate variability predict smoking outcomes. Front Hum Neurosci. 2012 Mar 19;6:54. doi: 10.3389/fnhum.2012.00054. eCollection 2012. PMID 22457646
- [Background] Koerten HR, Watford TS, Dubow EF, O'Brien WH. Cardiovascular effects of brief mindfulness meditation among perfectionists experiencing failure. Psychophysiology. 2020 Apr;57(4):e13517. doi: 10.1111/psyp.13517. Epub 2020 Feb 4. PMID 32020660